CLINICAL TRIAL: NCT01407991
Title: Placement of NG or OG Tube in Infants by Length Versus Traditional Measuring Methods
Brief Title: Nasogastric/Oral Gastric Tube Placement in Infants: Comparing 2 Measurement Methods
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study terminated due to change in clinical practice affecting recruitment. For majority of patients, NJ tubes are now used instead of NG tubes.
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 10-007863
Record Dates: First submitted 2011-07-25; First posted 2011-08-02 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Enteral Tube Placement
Keywords: Enteral tube placement

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Length or graph method (Experimental): The graph method is based on the infants' length determined by measurement using a length board and plotted on a graph derived from a formula to determine the depth for tube insertion (graph method). The graph method has been tested in the pediatric population but not in infants under six months of age (Klazner, Luke and Scalso, 2002). Using a graph method might reduce some of the variability in placement. We propose to extend the Klazner, Luke and Scalso (2002) study in the infant population.
  Interventions: Other: enteral tube placement accuracy
- NEM method for NG/OG tube placement (Active Comparator): Standard method- measure distance from the mouth to the ear and then the ear to mid abdomen and mark the tube to insert to that length. Nose to ear to mid-xiphoid-umbilicus (NEM).
  Interventions: Other: NEM method for NG/OG tube placement

INTERVENTIONS:
Other: enteral tube placement accuracy — The graph method is based on the infants' length determined by measurement using a length board and plotted on a graph derived from a formula to determine the depth for tube insertion (graph method). The graph method has been tested in the pediatric population but not in infants under six months of age (Klazner, Luke and Scalso, 2002). Using a graph method might reduce some of the variability in placement. We propose to extend the Klazner, Luke and Scalso (2002) study in the infant population.
  Arms: Length or graph method
Other: NEM method for NG/OG tube placement — measure distance from the mouth to the ear and then the ear to mid abdomen and mark the tube to insert to that length
  Arms: NEM method for NG/OG tube placement

SUMMARY:
The purpose of this study is to compare two methods of nasogastric/oral gastric (NG/OG) tube placement for efficacy and safety in the placement of NG/OG tube in infants less than 6 months of age. One method is based on the infant's length determined by measurement using a length board and plotted on a graph derived from a formula to determine the depth for tube insertion (graph method) and the other method is based on current standard of care, measuring from the nose to the ear and then the ear to mid abdomen (NEM) and mark the tube to know how far to insert the tube. Outcome comparison will be xray verification of placement.

DETAILED DESCRIPTION:
Preterm infants often require nutritional intake through a nasogastric or oral gastric tube to meet their high energy requirement and avoid aspiration of nutrition due to their immature suck/swallow reflex. When providing nutrition via an NG or OG tube, there are two basic safety issues; accurate placement, determined by the end of the tube reaching the mid abdominal area, and verification methods to assure placement is optimal. Based on a review of relevant literature, a potentially more accurate method of tube placement is available than the method used in current practice. We hypothesize the graph method will result in a more accurate and less variable placement of the NG tube into the mid-stomach of preterm infants than the current standard using the NEM method.

ELIGIBILITY:
Inclusion Criteria:

1. Infants less than 6 months of age in the neonatal intensive care unit (NICU) regardless of gestational age
2. Infants requiring an NG or OG tube for enteral feeds
3. Infants whose NG tube is placed by the bedside Registered Nurse (RN)
4. Parents need to speak and read English
5. Infant scheduled for X-Ray for standard of care (SOC) within 24hrs of scheduled NG/OG tube change or placement.

Exclusion Criteria:

1. Infants with congenital or structural anomalies of the GI tract
2. Infants with significant scoliosis
3. Infants with salem sump or repogle tube

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2011-07; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Evaluate safety and efficacy of Nasogastric/Orogastric tube placement using the length method | Participants will be followed for the duration of hospitalization, an average expected time of 4 weeks. Once an OG/NG tube change is completed per study protocol the participant will have completed the study.
  During the same day of NG/OG tube placement, verification of placement will be performed by bedside nurse as per institutional standards. X-ray verification will be done in batches (not same day) and read by radiologist blind to insertion method.

SECONDARY OUTCOMES:
compare depth ( too high, center, or too low) of NG/OG tube between the length method and the NEM method | X-ray outcome of NG/OG placement will be measured after every 10 subjects complete the study, on average 4 weeks.
  Radiologist blinded to the randomized method of insertion will determine location of placement.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Ely, PhD, RN, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Result] Klasner AE, Luke DA, Scalzo AJ. Pediatric orogastric and nasogastric tubes: a new formula evaluated. Ann Emerg Med. 2002 Mar;39(3):268-72. doi: 10.1067/mem.2002.120124. PMID 11867979